CLINICAL TRIAL: NCT04984512
Title: A Phase II/III ,Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled, Adaptive Design Study Evaluating the Efficacy And Safety of Mitizodone Phosphate Tablets in the Treatment of Patient With Major Depressive Disorder
Brief Title: The Efficacy And Safety Of Mitizodone Phosphate Tablets In The Treatment of Patient With Major Depressive Disorder
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC113995-P-5
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-07

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mitizodone Phosphate tablet 10mg (Experimental): Mitizodone Phosphate tablet 10mg ,orally,once daily for 8 weeks, then placebo,orally,once daily for 2 weeks.
  Interventions: Drug: Mitizodone Phosphate tablets
- Mitizodone Phosphate tablet 20mg (Experimental): Mitizodone Phosphate tablet 10mg ,orally,once daily for 1 weeks, then Mitizodone Phosphate tablet 20mg ,orally,once daily for 7 weeks, then Mitizodone Phosphate tablet 10mg ,orally,once daily for 1 weeks, then placebo,orally,once daily for 1 weeks.
  Interventions: Drug: Mitizodone Phosphate tablets
- Mitizodone Phosphate tablet 40mg (Experimental): Mitizodone Phosphate tablet 10mg ,orally,once daily for 1 weeks, then Mitizodone Phosphate tablet 20mg ,orally,once daily for 1 weeks, then Mitizodone Phosphate tablet 40mg ,orally,once daily for 6 weeks, then Mitizodone Phosphate tablet 20mg ,orally,once daily for 1 weeks, then Mitizodone Phosphate tablet 10mg ,orally,once daily for 1 weeks.
  Interventions: Drug: Mitizodone Phosphate tablets
- Placebo (Active Comparator): Placebo,tablet,orally,once daily for 10 weeks.
  Interventions: Drug: Placebo-matching tablets

INTERVENTIONS:
Drug: Mitizodone Phosphate tablets — Mitizodone Phosphate tablets will be administered with food.
  Other Names: HEC113995PA•H2O
  Arms: Mitizodone Phosphate tablet 10mg; Mitizodone Phosphate tablet 20mg; Mitizodone Phosphate tablet 40mg
Drug: Placebo-matching tablets — Placebo will be administered with food.
  Arms: Placebo

SUMMARY:
This is a phase 2 and 3 adaptive design study for Mitizodone Phosphate,to find out an optimal dose in phase 2 period and confirm the result an efficacy and safety in phase 3 period.Dose-finding will be done after 8 weeks of double-blinded treatment in phase 2 period and will be assessed by both efficacy and safety from 3 dose groups of Mitizodone Phosphate.The dose be found in phase 2 period will be evaluated on efficacy and safety when compared with placebo in phase 3 period with a duration of 8 weeks treatment.The target subjects are patients with MDD.

ELIGIBILITY:
Inclusion Criteria:

* 1.a Man or a woman with major depressive disorder(MDD) as the primary diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria (classification code 296.22、296.23、296.32、296.33)
* 2.Has a Montgomery Åsberg Depression Rating Scale (MADRS) total score of 26 or greater at Screening and Baseline Visits.
* 3.Has a Clinical Global Impression - Severity of Illness (CGI-S) score of 4 or greater at Screening and Baseline Visits.

Exclusion Criteria:

* 1.has major depressive disorder with psychotic features according to the DSM-5.
* 2.Current or history of: bipolar disorder、schizophrenia、anixety disorder、insomnia、any substance abuse or dependence and other psychiatry disorder as defined in the DSM-5.
* 3.Current or history of a clinically significant neurological disorder (including epilepsy、Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease).
* 4. has Serious body disease such as neurological disorders、cardiacvascular disorders、hepatic disorders、 renal disorders, blood system disorders and endocrine disorders.
* 5. Current or history of cancer( except basal cell of the skin and preinvasive carcinoma of cervix uteri).
* 6. Current or history of angle-closure glaucoma.
* 7. has made a suicide behavior in the previous 1 year ，or has a score greater than or equal to 4 on item 10 (suicidal thoughts) of MADRS .
* 8.has taken fluoxetine within 4 weeks prior to initial dosing.
* 9. has taken other antidepressive medications or antipsychotic medications within 2 weeks prior to initial dosing.
* 10.has psychotherap at Screening and/or Baseline Visits.
* 11.has had physiotherapy within 3 months prior to initial dosing.
* 12.Has an alanine aminotransferase, aspartate aminotransferase or total bilirubin level greater than 1.5 times the upper limits of normal.
* 13.Has an alanine aminotransferase, aspartate aminotransferase level greater than 2 times the upper limits of normal；or total bilirubin， direct bilirubin，creatinine level greater than 1.5 times the upper limits of normal；or a thyroid stimulating hormone value outside the normal range.
* 14.Has an abnormal electrocardiogram confirmed as clinically significant by the investigator.
* 15.Has a history of severe allergies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at week 8 | baseline and week 8
  The MADRS is a depression rating scale consisting of 10 items, each rated 0 (normal) to 6 (most abnormal). The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). A decrease in the total score or on individual items indicates improvement.

SECONDARY OUTCOMES:
Percentage of subjects With a MADRS Response at Week 8 | baseline and week 8
  Response is defined as a subject with a ≥50% decrease in Montgomery Åsberg Depression Rating Scale (MADRS) total score from Baseline.
Percentage of Participants in MADRS Remission at Week 8 | week 8
  Remission is defined as a participant with a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≤10.
Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at week 1、week 2 、week 4、week 6. | baseline 、 week 1、week 2 、week 4 and week 6.
  The MADRS is a depression rating scale consisting of 10 items, each rated 0 (normal) to 6 (most abnormal). The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). A decrease in the total score or on individual items indicates improvement.
Change From Baseline in the Clinical Global Impression - Severity of illness (CGI-S) Total Score at week 1、week 2 、week 4、week 6、week 8. | baseline、week 1、week 2 、week 4、week 6 and week 8.
  The Clinical Global Impression-Severity of illness scale assesses the subject's Severity as assessed by the clinician at the moment on a 8-point scale: 0, not assessed ; 1, normal，not at all ill ; 2, borderline mentally ill ; 3, mildly ill ; 4, moderately ill ; 5 , markedly ill ; 6, severely ill；7，among the most extremely ill patients.
Clinical Global Impression - Improvement (CGI-I) Score at week 1、week 2 、week 4、week 6、Week 8 | week 1、week 2 、week 4、week 6 and week 8.
  The Clinical Global Impression- Improvement scale assesses the subject's improvement (or worsening) as assessed by the clinician relative to Baseline on a 8-point scale: 0, not assessed ;1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Change From Baseline in the hamilton anxiety rating scale （HAM-A）Total Score at week 1、week 2 、week 4、week 6、week 8. | baseline、week 1、week 2 、week 4、week 6 and week 8.
  the HAM-A is a anxiety rating scale consisting of 14 items, each rated 0 (none) to 4 (very severe). The 14 items represent the core symptoms of anxiety illness. The overall score ranges from 0 (symptoms absent) to 56 (severe anxiety). A decrease in the total score or on individual items indicates improvement.

IPD SHARING:
Plan to Share IPD: No